CLINICAL TRIAL: NCT03556696
Title: Automatic Remifentanil Administration Guided by the Analgesia Nociception Index During Propofol Anesthesia
Brief Title: Automatic Remifentanil Administration Guided by ANI During Propofol Anesthesia
Acronym: ANI-LOOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016_48; 2017-A00858-45 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2018-04-10; First posted 2018-06-14 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-11

CONDITIONS: Nociceptive Pain; Surgical Procedure, Unspecified
Keywords: general anesthesia; analgesia/nociception balance monitoring; expert system
MeSH Terms: conditions — Nociceptive Pain; Agnosia | interventions — Remifentanil; Propofol

STUDY DESIGN:
Intervention Model Description: Monocentric prospective randomized controlled clinical trial
  * arm 1: medical device automatically administering remifentanil, guided by expert rules and continuous reading of heart rate, blood pressure and Analgesia Nociception Index (MDMS, Loos, France)
  * arm 2 : standard practice : remifentanil is administered using a target controlled device using a pK/pD model of Minto
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ANI-loop (Experimental): arm 1 : remifentanil is automatically administered by a medical device using expert rules and continuous reading of heart rate, blood pressure and Analgesia Nociception Index (MDMS, Loos, France)
  Interventions: Device: ANI-REMI-loop; Drug: Remifentanil; Drug: Propofol
- std_practice (Active Comparator): arm 2: remifentanil is administered by a target control device using Minto's remifentanil pK/pD model. This is standard practice for this type of surgery at the Burn Center of the University Hospital of Lille, France.
  Interventions: Device: remifentanil pK/pD target administration device; Drug: Remifentanil; Drug: Propofol; Device: ANI monitor

INTERVENTIONS:
Device: ANI-REMI-loop — experimental medical device using expert rules and continuous reading of heart rate, blood pressure and Analgesia Nociception Index for automatic remifentanil administration
  Arms: ANI-loop
Device: remifentanil pK/pD target administration device — standard practice, remifentanil administration using Minto's pK/pD model
  Arms: std_practice
Drug: Remifentanil — Remifentanil Ce target can range from 0 to 10 ng.ml-1. Remifentanil target is adapted in order to maintain Analgesia Nociception Index (MDMS, Loos, France) in the [50-70] range.
Drug: Propofol — propofol is used for induction and maintenance of general anesthesia using Schnider pK/pD model. Propofol Ce target is adapted in order to maintain BiSpectral Index in [40-60] range
Device: ANI monitor — ANI (Analgesia Nociception Index) value is used in the "std_practice" arm for guidance of the remifentanil Ce target
  Other Names: PhysioDoloris (MDMS, Loos, France)
  Arms: std_practice

SUMMARY:
Prospective Randomized Monocentric Clinical Trial during propofol anesthesia. The aim of the study is to test whether the use of a medical device designed to automatically administer remifentanil during surgery based on expert rules and continuous reading of heart rate, blood pressure and the Analgesia Nociception Index results in lower overall remifentanil administration versus standard practice.

DETAILED DESCRIPTION:
Prospective Randomized Monocentric Clinical Trial during propofol anesthesia.

* inclusion: ASA 1, 2 or 3 adult patients scheduled to undergo burn wound surgery in a Burn Center (University Hospital of Lille, France)
* arm 1 : Remifentanil will be automatically administered by an expert system guided by heart rate, blood pressure and the Analgesia Nociception Index (ANI).
* arm 2 : Remifentanil will be administered by a target controlled device using the Minto pK/pD model.
* propofol is administered throughout the procedure with a target controlled device using the pK/pD model of Schnider. The target will be guided by the BiSpectral index values.
* primary endpoint : overall normalized remifentanil administration.
* secondary endpoints : relative amount of time spent in a state of hemodynamic reactivity ; relative amount of time the ANI spends in the [0-50], [50-70] and [70-100] windows ; relative amount of time the BIS spends in the [0-40], [40-60] and [60-100] ; hemodynamic status at various times during anesthesia ; total amount of target modifications of remifentanil and propofol ; total amount of morphine administered in PACU ; total amount of ketamine administered in PACU ; incidence of nausea/vomiting in PACU ;

ELIGIBILITY:
Inclusion Criteria:

* ASA 1, 2 or 3 adult patients scheduled to undergo burn wound surgery at the Burn Center of the University Hospital of Lille

Exclusion Criteria:

* BMI outside [17 - 35 kg/m2]
* pregnancy or breast feeding women
* non sinus cardiac rhythm
* documented dysautonomia
* complicated diabetes mellitus
* known allergy to a drug used in the clinical trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2018-06-27 (Actual); Primary Completion 2022-06-14 (Actual); Study Completion 2022-11-22 (Actual)

PRIMARY OUTCOMES:
normalized remifentanil administration | During the surgery, an average Three hours and a half
  ratio of total amount of administered remifentanil with body weight and duration of administration

SECONDARY OUTCOMES:
hemodynamic reactivity or bradycardia or hypotension | During the surgery, an average Three hours and a half
  relative amount of time during which heart rate or SBP exceed 120% of baseline, or heart rate drops below 40/min, or SBP drops below 75 mmHg.
total administered ephedrine | duration of general anesthesia
  total amount of ephedrine administered during general anesthesia
Analgesia Nociception Index (ANI) | During the surgery, an average Three hours and a half
  relative amount of time spent with ANIi in the [0-50], [50-70] and [70-100] windows. Same with ANIm
Bispectral Index (BIS) | During the surgery, an average Three hours and a half
  relative amount of time spent with BIS in the [0-40], [40-60] and [60-100] windows.
Change antinociception/nociception balance status | 5 min before start of nociception, 5 min after start of nociception and 20 min after start of nociception
  composite measure: heart rate, blood pressure, ANIi, ANIm, end-tidal CO2, PeakPressure
Pain in PACU | During the first two postoperative hours
  Visual Analog Scale every 15 min in PACU The pain VAS is a continuous scale comprised of a horizontal (HVAS) or vertical (VVAS) line, usually 10 centimeters (100 mm) in length, anchored by 2 verbal descriptors, one for each symptom extreme (0, 10).
morphine in PACU | During the first two postoperative hours
  Total amount of administered morphine during PACU stay
ketamine in PACU | During the first two postoperative hours
  Total amount of administered ketamine during PACU stay
nausea/vomiting in PACU | During the first two postoperative hours
  reported number of nausea/vomiting during PACU stay
remi target changes | During the surgery, an average Three hours and a half
  total number of target changes during general anesthesia
propofol target changes | During the surgery, an average Three hours and a half
  total number of target changes during general anesthesia
normalized propofol administration | During the surgery, an average Three hours and a half
  ratio of total amount of propofol administered with body weight and duration of general anesthesia
ANI-REMI-loop switch to manual | During the surgery, an average Three hours and a half
  number of interventions on ANI-REMI-loop device: switch to manual

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu JEANNE, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Roger Salengro, CHU, Lille, France